CLINICAL TRIAL: NCT04451005
Title: Development of a New Sarcopenia Screening Tool in the Elderly
Brief Title: Diagnostic Evaluation of Sarcopenia in Elderly Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Dan Linetzky Waitzberg, Principal researcher, University of Sao Paulo
Other Study IDs: SARC-F
Record Dates: First submitted 2020-06-02; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Sarcopenia
Keywords: Body composition; Sarcopenia; Elderly
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly patients with sarcopenia: Elderly patients with sarcopenia
  Interventions: Other: 0

INTERVENTIONS:
Other: 0 — Elderly patients with sarcopenia

SUMMARY:
Sarcopenia is a generalized progressive skeletal muscle disorder that represents a related physiological vulnerability that is associated with or increases the likelihood of adverse outcomes, including falls, fractures, physical disability and death. The parameters used to assess sarcopenia in clinical practice have limited use due to their custody.

In this perspective, this study proposes or develops a tool for the diagnosis of having sarcopenia with a specific boa and a sensitive boa.

low cost and useful.

Elderly patients (n = 403) from the Geriatrics Outpatient Clinic of Hospital das Clínicas, Faculty of Medicine, University of São Paulo will be selected

This study was of clinical importance, due to sarcopenia and a relevant factor, and could lead to consequences and poor prognosis in patients with gold, and it was not a method of clinical practice to properly endorse body composition in this population.

DETAILED DESCRIPTION:
Sarcopenia is a progressive and generalized skeletal muscle disorder that represents an age-related physiological vulnerability that is associated with an increased likelihood of adverse outcomes, including falls, fractures, physical disability and mortality. The parameters used to assess sarcopenia in clinical practice have limited use due to its cost.

In this perspective, this study proposes the development of a tool for the diagnosis of having sarcopenia with good specificity and good sensitivity and of low cost and useful.

Elderly patients (n = 403) from the Geriatrics Outpatient Clinic of Hospital das Clínicas, Faculty of Medicine, University of São Paulo will be selected. After signing the informed consent, sarcopenia will be assessed using the reference method (DXA) and anthropometry. The data obtained by the methods are treated statistically to obtain correlation and thus a new tool for the evaluation of sarcopenia patients in the elderly can be developed.

This study is of clinical importance, as sarcopenia is a relevant factor and can lead to consequences and poor prognosis in elderly patients, and there is no low-cost method in clinical practice to properly assess body composition in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Sign free and informed consent;
* Demonstrate interest, conditions and availability to participate in all procedures included in the study protocol;

Exclusion Criteria:

* Refusal to participate;
* Patients who have not undergone cognitive testing;
* Physical amputation;
* Patients undergoing interventional treatment for sarcopenia;

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly patients over 60 years old, with cognitive ability and interested in participating in the study
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Sarcopenia in the elderly | 12 months
  Evaluation of sarcopenia in the elderly

SECONDARY OUTCOMES:
Development of a new tool for sarcopenia screening | 12 months
  Development of a new tool for sarcopenia screening